CLINICAL TRIAL: NCT00312208
Title: A Multicenter Phase III Randomized Trial Comparing Docetaxel in Combination With Doxorubicin and Cyclophosphamide Versus Doxorubicin and Cyclophosphamide Followed by Docetaxel as Adjuvant Treatment of Operable Breast Cancer HER2neu Negative Patients With Positive Axillary Lymph Nodes
Brief Title: Docetaxel in Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Cancer International Research Group (CIRG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAX_GMA_301; BCIRG 005
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Results first posted 2010-02-17 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Cyclophosphamide

ARMS (2):
- 1 (Experimental): Doxorubicin in combination with cyclophosphamide followed by docetaxel (AC -> T)
  Interventions: Drug: Docetaxel,doxorubicin, cyclophosphamide
- 2 (Experimental): Docetaxel in combination with doxorubicin and cyclophosphamide (TAC)
  Interventions: Drug: docetaxel, doxorubicin, cyclophosphamide

INTERVENTIONS:
Drug: docetaxel, doxorubicin, cyclophosphamide — TAC x 6 : Docetaxel 75 mg/m² as 1 hour IV infusion on day 1 every 3 weeks in combination with doxorubicin 50 mg/m² as an IV bolus and cyclophosphamide 500 mg/m2 as IV on day 1 every 3 weeks. Sequence of administration is as follows: doxorubicin followed by cyclophosphamide followed by docetaxel.
  Arms: 2
Drug: Docetaxel,doxorubicin, cyclophosphamide — AC x 4: Doxorubicin 60 mg/m² as an IV bolus in combination with cyclophosphamide 600 mg/m² as IV followed by docetaxel 100 mg/m² as 1 hour IV infusion on day 1 every 3 weeks for 4 cycles.
  Arms: 1

SUMMARY:
Primary objective :

* To compare disease-free survival after treatment with docetaxel in combination with doxorubicin and cyclophosphamide to doxorubicin and cyclophosphamide followed by docetaxel in operable adjuvant breast cancer HER2neu negative patients with positive axillary lymph nodes.

Secondary objectives :

* To compare toxicity and quality of life between the 2 above-mentioned arms.
* To evaluate pathologic and molecular markers for predicting efficacy.

ELIGIBILITY:
Inclusion Criteria :

* Histologically proven breast cancer. Interval between definitive surgery that includes axillary lymph node dissection and registration is less than or equal to 60 days. A central pathology review may be performed post randomization for confirmation of diagnosis and molecular studies.
* Definitive surgical treatment must be either mastectomy, or breast conserving surgery with axillary lymph node dissection for operable breast cancer (T1-3, Clinical N0-1, M0). Margins of resected specimen from definitive surgery must be histologically free of invasive adenocarcinoma and Ductal Carcinoma In Situ (DCIS). Lobular carcinoma in-situ does not count as a positive margin.
* Histologic examination of the tumor: Invasive adenocarcinoma with at least one axillary lymph node (pN1) showing evidence of tumor among a minimum of six resected lymph nodes.
* Tumor must show negative HER2 neu proto-oncogene overexpression by FISH (Fluorescence In Situ Hybridization). Confirmation of non overexpression will be centrally assessed by authorized BCIRG (Breast Cancer International Research Group) laboratories prior to randomization.
* Estrogen and/or progesterone receptor analysis performed on the primary tumor prior to randomization. Results must be known at the time of randomization.(Note: Patients whose tumor is estrogen receptor negative with progesterone receptor status unknown or undetermined, must have the progesterone receptor assayed in order to determine hormonal receptor status. Patients whose tumor is progesterone receptor negative with estrogen receptor status unknown or undetermined, must have the estrogen receptor assayed in order to determine hormonal receptor status).
* Karnofsky Performance status index > 80%.
* Normal cardiac function must be confirmed by LVEF (Lef Ventricular Ejection Fraction) i.e. MUGA (Multi Gated Acquisition) scan or echocardiography and ECG within 3 months prior to registration. LVEF result must be above or equal to the lower limit of normal for the institution. The ECG results must be within normal limits or show no significant abnormalities.
* Laboratory requirements: (within 14 days prior to registration)

  * Hematology:

    * Neutrophils > or = 2.0 x 10^9/L
    * Platelets > or = 100 x 10^9/L
    * Hemoglobin > or = 10 g/dL
  * Hepatic function:

    * Total bilirubin < or = 1 UNL (Upper Normal Limit)
    * ASAT (Aspartate Amino Transferase) and ALAT (Alanine Amino Transferase) < or = 2.5 UNL
    * Alkaline phosphatase < or = 5 UNL
    * Patients with ASAT and/or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study.
  * Renal function:

    * Creatinine < or = 175 µmol/L (2 mg/dL);
    * If limit reached, the calculated creatinine clearance should be > or = 60mL/min.
* Complete staging work-up within 3 months prior to registration. All patients will have contralateral mammography, chest X-ray (Posteroanterior and lateral) and/or CT scan and/or MRI (Magnetic Resonance Imaging), abdominal ultrasound and/or CT scan (computerized tomography) and/or MRI, and bone scan. In case of positive bone scan, bone X-ray is mandatory to rule out the possibility of non-metastatic hot spots. Other tests may be performed as clinically indicated.
* Negative pregnancy test (urine or serum) within 7 days prior to registration for all women of childbearing potential.

Exclusion Criteria :

* Prior systemic anticancer therapy for breast cancer (immunotherapy, hormonotherapy, genetherapy , chemotherapy).
* Prior anthracycline therapy or taxoids (paclitaxel, docetaxel) for any malignancy.
* Prior radiation therapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant, or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures during study treatment (chemotherapy and tamoxifen therapy) and must have negative urine or serum pregnancy test within 7 days prior to registration.
* Any T4 or N2 or known N3 or M1 breast cancer.
* Pre-existing motor or sensory neurotoxicity of a severity > grade 2 by NCI-CTC (National Cancer Institute - Common Toxicity Criteria), version 2.0.
* Other serious illness or medical condition:

  * congestive heart failure or unstable angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or high-risk uncontrolled arrhythmias
  * history of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
  * active uncontrolled infection
  * active peptic ulcer, unstable diabetes mellitus
* Past or current history of neoplasm other than breast carcinoma, except for:

  * curatively treated non-melanoma skin cancer
  * carcinoma in situ of the cervix
  * other cancer curatively treated and with no evidence of disease for at least 10 years
  * ipsilateral ductal carcinoma in-situ (DCIS) of the breast
  * lobular carcinoma in-situ (LCIS) of the breast
* Chronic treatment with corticosteroids unless initiated > 6 months prior to study entry and at low dose (< 20 mg methylprednisolone or equivalent).
* Concurrent treatment with ovarian hormonal replacement therapy. Prior treatment should be stopped before study entry.
* Definite contraindications for the use of corticosteroids.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
* Concurrent treatment with any other anti-cancer therapy.
* Current therapy with any hormonal agent such as raloxifene, tamoxifen or other selective estrogen receptor modulators (SERMs), either for osteoporosis or prevention. Patients must have discontinued these agents prior to randomization.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3299 (Actual)
Dates: Start 2001-11; Primary Completion 2008-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe AUSSEL, Study Director — Sanofi
Locations (37):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Buenos Aires, Argentina
- Sanofi-Aventis, Macquarie Park, Australia
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, Sarajevo, Bosnia and Herzegovina
- Sanofi-Aventis, São Paulo, Brazil
- Sanofi-Aventis, Sofia, Bulgaria
- Sanofi-Aventis, Laval, Canada
- Sanofi-Aventis, Shanghai, China
- Sanofi-Aventis, Bogotá, Colombia
- Sanofi-Aventis, Zagreb, Croatia
- Sanofi-Aventis, Nicosia, Cyprus
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Cairo, Egypt
- Sanofi-Aventis, Tallinn, Estonia
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Kallithea, Greece
- Sanofi-Aventis, Hong Kong, Hong Kong
- Sanofi-Aventis, Budapest, Hungary
- Sanofi-Aventis, Dublin, Ireland
- Sanofi-Aventis, Netanya, Israel
- Sanofi-Aventis, Beirut, Lebanon
- Sanofi-Aventis, México, Mexico
- Sanofi-aventis, Auckland, New Zealand
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Porto Salvo, Portugal
- Sanofi-Aventis, Bucharest, Romania
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Jeddah, Saudi Arabia
- Sanofi-Aventis, Ljubljana, Slovenia
- Sanofi-Aventis, Midrand, South Africa
- Sanofi-Aventis, Seoul, South Korea
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Taipei, Taiwan
- Sanofi-Aventis, Montevideo, Uruguay
- Sanofi-Aventis, Caracas, Venezuela

REFERENCES:
- [Derived] Blasco A, Lopez-Tarruella S, Urruticoechea A, Carrasco E, Spera G, Martin M, Bermejo B, Chap L, Ruiz-Borrego M, Crown J, Garcia-Saenz JA, Chan A, Guerrero-Zotano A, Semiglazov V, Calvo L, Pienkowski T, Herranz J, Slamon D. Intermediate endpoints as surrogates for long-term outcomes in breast cancer adjuvant chemotherapy trials. Oncologist. 2025 Sep 1;30(9):oyaf263. doi: 10.1093/oncolo/oyaf263. PMID 40838872
- [Derived] Press MF, Sauter G, Buyse M, Fourmanoir H, Quinaux E, Tsao-Wei DD, Eiermann W, Robert N, Pienkowski T, Crown J, Martin M, Valero V, Mackey JR, Bee V, Ma Y, Villalobos I, Campeau A, Mirlacher M, Lindsay MA, Slamon DJ. HER2 Gene Amplification Testing by Fluorescent In Situ Hybridization (FISH): Comparison of the ASCO-College of American Pathologists Guidelines With FISH Scores Used for Enrollment in Breast Cancer International Research Group Clinical Trials. J Clin Oncol. 2016 Oct 10;34(29):3518-3528. doi: 10.1200/JCO.2016.66.6693. PMID 27573653
- [Derived] Mackey JR, Pienkowski T, Crown J, Sadeghi S, Martin M, Chan A, Saleh M, Sehdev S, Provencher L, Semiglazov V, Press MF, Sauter G, Lindsay M, Houe V, Buyse M, Drevot P, Hitier S, Bensfia S, Eiermann W. Long-term outcomes after adjuvant treatment of sequential versus combination docetaxel with doxorubicin and cyclophosphamide in node-positive breast cancer: BCIRG-005 randomized trial. Ann Oncol. 2016 Jun;27(6):1041-1047. doi: 10.1093/annonc/mdw098. Epub 2016 Mar 2. PMID 26940688

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T): AC x 4: Doxorubicin 60 mg/m² as an IV bolus in combination with cyclophosphamide 600 mg/m² as IV followed by docetaxel 100 mg/m² as 1 hour IV infusion on day 1 every 3 weeks for 4 cycles.
- Docetaxel + Doxorubicin and Cyclophosphamide (TAC): TAC x 6 : Docetaxel 75 mg/m² as 1 hour IV infusion on day 1 every 3 weeks in combination with doxorubicin 50 mg/m² as an IV bolus and cyclophosphamide 500 mg/m2 as IV on day 1 every 3 weeks. Sequence of administration is as follows: doxorubicin followed by cyclophosphamide followed by docetaxel.
Period: Overall Study
Arm/Group | Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T) | Docetaxel + Doxorubicin and Cyclophosphamide (TAC)
Started | 1649 (1649 patients randomized, 1634 patients treated) | 1649 (1649 patients randomized 1635 patients treated)
Completed | 1477 | 1526
Not Completed | 172 | 123
Not completed — Adverse Event | 97 | 61
Not completed — Protocol Violation | 5 | 3
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 7 | 4
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 53 | 42
Not completed — Other | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T) | Docetaxel + Doxorubicin and Cyclophosphamide (TAC) | Total
Number analyzed (Participants) | 1649 | 1649 | 3298
Age, Customized [Number; unit: Participants]
  > =65 years | 85 | 83 | 168
  Between 65 and 50 years | 784 | 783 | 1567
  Between 49 and 35 years | 689 | 710 | 1399
  < =35 years | 91 | 73 | 164
Age, Continuous [Median (Full Range); unit: years] | 50 [22 to 74] | 50 [24 to 72] | 50 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1649 | 1649 | 3298
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 31 | 32 | 63
  Australia | 156 | 144 | 300
  Belgium | 33 | 31 | 64
  Bosnia And Herzegovina | 5 | 5 | 10
  Brazil | 19 | 21 | 40
  Bulgaria | 11 | 11 | 22
  Canada | 174 | 180 | 354
  China | 21 | 17 | 38
  Colombia | 6 | 8 | 14
  Croatia | 29 | 29 | 58
  Cyprus | 2 | 5 | 7
  Czech Republic | 11 | 10 | 21
  Egypt | 4 | 4 | 8
  Estonia | 3 | 2 | 5
  France | 59 | 58 | 117
  Germany | 224 | 223 | 447
  Greece | 5 | 3 | 8
  Hong Kong | 3 | 6 | 9
  Hungary | 34 | 35 | 69
  Ireland | 83 | 88 | 171
  Israel | 63 | 67 | 130
  Lebanon | 23 | 18 | 41
  Mexico | 5 | 3 | 8
  New Zealand | 21 | 19 | 40
  Poland | 167 | 168 | 335
  Portugal | 2 | 1 | 3
  Russian Federation | 32 | 35 | 67
  Romania | 17 | 19 | 36
  Saudi Arabia | 2 | 0 | 2
  Slovenia | 15 | 17 | 32
  South Africa | 19 | 21 | 40
  South Korea | 22 | 27 | 49
  Spain | 26 | 41 | 67
  Taiwan | 18 | 16 | 34
  United States | 294 | 278 | 572
  Uruguay | 4 | 2 | 6
  Venezuela | 6 | 5 | 11
Hormonal Receptor Status [Number; unit: Participants]
  Positive | 1348 | 1346 | 2694
  Negative | 301 | 303 | 604
Karnofsky Performance Status at Baseline [Number; unit: Participants]
  80 - Activity with effort; some signs of disease | 36 | 33 | 69
  90 - Normal activity; minor signs of disease | 315 | 323 | 638
  100 - Normal no complaints; no evidence of disease | 1298 | 1293 | 2591
Menopausal status [Number; unit: Participants]
  Pre-Menopausal or Other age < 50 Years | 866 | 863 | 1729
  Post-Menopausal or Other age > 50 Years | 783 | 786 | 1569
Number of Positive Lymph Nodes [Number; unit: Participants]
  [0] | 0 | 1 | 1
  [1 to 3] | 1010 | 1005 | 2015
  [4 to 10] | 462 | 456 | 918
  > 10 | 177 | 187 | 364
Patients with at least one surgery [Number; unit: Participants]
  Mastectomy | 955 | 973 | 1928
  Lumpectomy | 283 | 276 | 559
  Quadrantectomy/Segmental | 411 | 400 | 811
Primary Tumor [Number; unit: Participants]
  pT1: Tumor < = 2cm | 692 | 668 | 1360
  pT2: Tumor in [ 2 - 5 ] | 824 | 844 | 1668
  pT3: Tumor > 5cm | 131 | 135 | 266
  pT4: Tumor with extension to chest wall/skin | 1 | 2 | 3
  pTis: Carcinoma in situ | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Local, Regional or Metastatic Relapse, or Second Primary Cancer, or Death From Any Cause (Disease-Free Survival)
Description: The primary event is the local, regional or metastatic relapse or the date of second primary cancer or death from any cause (whichever occurs first). The primary efficacy analysis is performed on the time from randomization to this primary event. The Measured Values table below presents the numbers of patients with the event at the end of the study period.
Time Frame: Median follow-up 65 months
Population: The primary efficacy analysis was performed on the Intent-to-Treat (ITT) population. Although the original Outcome Measure was intended to be presented as median disease free survival time, median time-to-event was not reached in any group; therefore, number of participants with relapse was presented.
Measure: Number; unit: Participants
Arm/Group | Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T) | Docetaxel + Doxorubicin and Cyclophosphamide (TAC)
Number analyzed (Participants) | 1649 | 1649
Participants | 356 | 352
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T) vs Docetaxel + Doxorubicin and Cyclophosphamide (TAC); Test type: Superiority or Other; p = 0.978, Log Rank — Cumulative incidence functions in each treatment group were calculated using non-parametric Kaplan-Meier estimates; Hazard Ratio (HR) = 1.00, 95% CI [0.86 to 1.16]

2. Secondary Outcome: Death From Any Cause (Overall Survival)
Description: The considered event is death from any cause. The analysis is performed on the time from randomization to this event. The Measured Values table below presents the numbers of patients with the event at the end of the study period.
Time Frame: Median follow-up of 65 months
Population: The analysis was performed on the Intent-to-Treat (ITT) population. Although the original Outcome Measure was intended to be presented as median survival time, median time-to-event was not reached in any group; therefore, number of participants who died was presented.
Measure: Number; unit: Participants
Arm/Group | Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T) | Docetaxel + Doxorubicin and Cyclophosphamide (TAC)
Number analyzed (Participants) | 1649 | 1649
Participants | 187 [65.64 to 65.91] | 202 [65.48 to 65.84]
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T) vs Docetaxel + Doxorubicin and Cyclophosphamide (TAC); Test type: Superiority or Other; p = 0.371, Log Rank — Cumulative incidences calculated in each group using non-parametric Kaplan-Meier estimates; Hazard Ratio (HR) = 0.91, 95% CI [0.75 to 1.11]

ADVERSE EVENTS:
Description: The number of patients at risk corresponds to the patients who received at least one dose of treatment
Arm/Group | Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T) | Docetaxel + Doxorubicin and Cyclophosphamide (TAC)
Serious Adverse Events (participants affected / at risk) | 331/1634 | 520/1635
Other Adverse Events (participants affected / at risk) | 1634/1634 | 1629/1635
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T) (N=1634) | Docetaxel + Doxorubicin and Cyclophosphamide (TAC) (N=1635)
Abdominal Syndrom Acute (General disorders) | 1 | 0
Allergic Reaction (General disorders) | 7 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Anemia (Blood and lymphatic system disorders) | 3 | 5
Anorexia (Gastrointestinal disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 3 | 3
Arrhythmia Ventricular (Cardiac disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Asthenia (General disorders) | 5 | 5
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cellulitis (General disorders) | 6 | 1
Cerebrovascular Accident (Vascular disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 0
Coagulation disorders (Blood and lymphatic system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 1 | 8
Convulsion (Nervous system disorders) | 1 | 2
Creatinine increase (Renal and urinary disorders) | 0 | 2
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cystitis (Renal and urinary disorders) | 0 | 2
Deaf (Ear and labyrinth disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 6
Delusions (Nervous system disorders) | 1 | 0
Depression (Nervous system disorders) | 2 | 1
Derm Exfoliating (Skin and subcutaneous tissue disorders) | 8 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 13 | 13
Dizziness (Nervous system disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Edema (Metabolism and nutrition disorders) | 0 | 1
Edema Peripheral (Metabolism and nutrition disorders) | 5 | 1
Effusion Pericardial (Cardiac disorders) | 1 | 0
Effusion Pleural (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emotional Lability (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Erythema Multiform (Skin and subcutaneous tissue disorders) | 1 | 0
Fever (including serious febrile neutropenia) (General disorders) | 122 | 293
Fibrillation Ventricular (Cardiac disorders) | 0 | 1
Fibrosis lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastro-intestinal Disorder (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 2
Headache (General disorders) | 1 | 1
Heart Arrest (Cardiac disorders) | 1 | 0
Heart Failure Left (Cardiac disorders) | 3 | 0
Hemorrhage Intracranial (Vascular disorders) | 1 | 0
Hemorrhage Rectal (Gastrointestinal disorders) | 2 | 1
Hemorrhage Retinal (Eye disorders) | 0 | 1
Hemorrhage Vaginal (Blood and lymphatic system disorders) | 1 | 0
Herpes Zoster (Skin and subcutaneous tissue disorders) | 1 | 0
Hydrocephalus (General disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Cardiac disorders) | 4 | 3
Ileus (Gastrointestinal disorders) | 1 | 1
Infection (including neutropenic infection) (Infections and infestations) | 86 | 143
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 | 1
Injury Accident (Injury, poisoning and procedural complications) | 3 | 0
Ischemia myocardial (Cardiac disorders) | 0 | 2
Kidney Failure (Renal and urinary disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 18 | 56
Liver Failure (Hepatobiliary disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphedema (Blood and lymphatic system disorders) | 0 | 2
Mastitis (Renal and urinary disorders) | 0 | 1
Melena (Gastrointestinal disorders) | 0 | 1
Menstrual Disorder (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Mucous Membrane Disorder (General disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 14 | 19
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm Uterine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 6 | 3
Nodule skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pain (General disorders) | 3 | 1
Pain Abdominal (General disorders) | 1 | 3
Pain Biliary (General disorders) | 1 | 0
Pain Chest (General disorders) | 3 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Papilledema (Eye disorders) | 1 | 0
Paralysis Vocal Cord (Nervous system disorders) | 0 | 1
Peritonitis (General disorders) | 0 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Interstitial (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pregnancy Unintended (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Proctitis (Gastrointestinal disorders) | 1 | 1
Psychosis (Psychiatric disorders) | 1 | 0
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
SGOT Increase (Hepatobiliary disorders) | 2 | 0
SGPT Increase (Hepatobiliary disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 8 | 9
Syncope (Cardiac disorders) | 8 | 5
Tachycardia (Cardiac disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombophlebitis Deep (Vascular disorders) | 14 | 14
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Ulcer Stomach (Gastrointestinal disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1
Urinary Tract Disorder (Renal and urinary disorders) | 0 | 1
Uterine Fibroid Enlargement (Reproductive system and breast disorders) | 1 | 0
Vaginitis (Reproductive system and breast disorders) | 0 | 1
Vertigo (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 16 | 28
Vulvovaginitis (Reproductive system and breast disorders) | 1 | 0
Weight Increase (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin + Cyclophosphamide Followed by Docetaxel (AC -> T) (N=1634) | Docetaxel + Doxorubicin and Cyclophosphamide (TAC) (N=1635)
Allergic reaction (General disorders) | 172 | 190
Alopecia (Skin and subcutaneous tissue disorders) | 1601 | 1587
Anemia (Blood and lymphatic system disorders) | 461 | 658 — NCI severity grade was derived based on reported laboratory data
Anorexia (Gastrointestinal disorders) | 370 | 376
Arthralgia (Musculoskeletal and connective tissue disorders) | 602 | 382
Asthenia (Musculoskeletal and connective tissue disorders) | 1328 | 1310
Conjunctivitis (Eye disorders) | 176 | 131
Constipation (Gastrointestinal disorders) | 599 | 555
Cough (Respiratory, thoracic and mediastinal disorders) | 211 | 222
Depression (Nervous system disorders) | 160 | 132
Derm exfoliating (Skin and subcutaneous tissue disorders) | 143 | 36
Diarrhea (Gastrointestinal disorders) | 644 | 606
Dizziness (Nervous system disorders) | 149 | 169
Dry eye (Eye disorders) | 87 | 65
Dry mouth (Nervous system disorders) | 149 | 80
Dyspepsia (Gastrointestinal disorders) | 339 | 387
Dysphagia (Gastrointestinal disorders) | 83 | 65
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 319 | 287
Edema peripheral (Metabolism and nutrition disorders) | 488 | 417
Emotion labil (Nervous system disorders) | 168 | 111
Epistaxis (Blood and lymphatic system disorders) | 123 | 72
Fever (including febrile neutropenia) (General disorders) | 289 | 467
Headache (General disorders) | 433 | 370
Infection (including neutropenic infection) (Infections and infestations) | 573 | 457
Injection site reaction (General disorders) | 124 | 92
Insomnia (Nervous system disorders) | 334 | 277
Lacrimation disorder (Eye disorders) | 357 | 212
Leucopenia (Blood and lymphatic system disorders) | 59 | 88
Lymphedema (Blood and lymphatic system disorders) | 101 | 109
Menses disorder (Reproductive system and breast disorders) | 489 | 501
Myalgia (Musculoskeletal and connective tissue disorders) | 834 | 587
Nail disorder (Skin and subcutaneous tissue disorders) | 729 | 363
Nausea (Gastrointestinal disorders) | 1435 | 1334
Neuropathy (Nervous system disorders) | 723 | 482
Neutropenia (Blood and lymphatic system disorders) | 1133 | 1049 — NCI severity grade was derived based on reported laboratory data
Pain (General disorders) | 275 | 235
Pain abdominal (General disorders) | 256 | 271
Pain back (General disorders) | 123 | 121
Pain bone (General disorders) | 230 | 204
Pain chest (General disorders) | 93 | 76
Palpitations (Cardiac disorders) | 82 | 84
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 88 | 69
Proctitis (Gastrointestinal disorders) | 82 | 100
Rash maculopapular (Skin and subcutaneous tissue disorders) | 402 | 314
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 268 | 198
Skin dry (Skin and subcutaneous tissue disorders) | 107 | 85
Stomatitis (Gastrointestinal disorders) | 1035 | 1026
Sweating (Skin and subcutaneous tissue disorders) | 77 | 93
Taste pervers (Gastrointestinal disorders) | 480 | 426
Thrombocytopenia (Blood and lymphatic system disorders) | 52 | 109 — NCI severity grade was derived based on reported laboratory data
Vasodilatation (Nervous system disorders) | 388 | 437
Vomiting (Gastrointestinal disorders) | 907 | 742
Weight decrease (General disorders) | 116 | 140
Weight increase (General disorders) | 370 | 240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.